CLINICAL TRIAL: NCT03373279
Title: Bioelectrical Impedance Spectroscopy in Heart Transplantation: Tracking Post-Transplant Changes in Body Composition and Correlation With Conventional Preoperative Risk Assessment Modalities
Acronym: BIS
Status: Completed | Type: Observational
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 016-114
Record Dates: First submitted 2017-12-05; First posted 2017-12-14 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2023-01

CONDITIONS: Heart Transplant Failure and Rejection
Keywords: Heart Transplant
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with marginal physiologic reserve, severe frailty, and/or malnutrition may be regarded as unsuitable candidates for advanced cardiac replacement therapies. However, little data exist on precisely which measures are predictive of subsequent adverse events. Assessment of nutritional status and frailty is still largely predicated on crude and obsolete parameters, such as baseline serum albumin level or body mass index (BMI). In this prospective cohort study the investigators will evaluate the use of bio-electrical impedance spectroscopy (BIS) as a measure of body composition and assess the associations with surgical outcomes.

DETAILED DESCRIPTION:
This is a prospective cohort study, with study visits at Enrollment and subsequently at ≤10 days , 1 month (+/- 7 days), 3 months (+/- 7 days) , 6 months (+/- 14 days) , and 12 months (+/- 14 days) after heart transplant surgery.

BIS measurements will be performed on patients both in the pretransplant and post-transplant periods except when contraindicated in the pretransplant setting concerning patients with advanced heart failure. Because the use of BIS is contraindicated in the setting of permanent pacemaker and/or internal cardiac defibrillator (ICD) devices, BIS assessment cannot be performed in the pretransplant setting for patients with advanced heart failure as the majority of these patients already have these devices in place. However, at the time of cardiac transplantation, these devices will be removed from those patients with advanced heart failure and the BIS measurements will then be performed shortly after transplantation, and then serially during the post-transplant period at various time intervals for one year in order to track changes in body composition.

These measurements will be compared to traditional measurements performed at the time of preoperative evaluation by the nutritional and dietitian support team.

ELIGIBILITY:
Inclusion Criteria:

* Listed for a native heart transplant at BUMC
* At least 18 years of age

Exclusion Criteria:

* Women during pregnancy
* Patient currently has a ventricular assist device

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving a heart transplant
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
BIS Parameters Predictive of Adverse Outcomes | 5 years
  BIS-derived elements such as FM and FFM will be compared with standard preoperative variables for correlation of malnutrition assessment and predictability of adverse clinical events such as mortality, primary graft dysfunction, rejection, acute kidney injury, prolonged hospital stay, and hospital readmission. Several measures of nutrition status will be measured including SGA, BMI, tricep skinfolds, midarm muscle circumference, and FFM via BIS. The methods will be compared to determine agreement among the methods in determining malnutrition. In addition, nutrition status measures will be repeated at specified times over the first year following heart transplantation to describe the changes in body composition after transplantation. These changes occur gradually and thus the initial postoperative measurement will be closely representative of the patient's initial (pre-transplant) baseline status.

CONTACTS AND LOCATIONS:
Overall Officials: Jeaette Hasse, RD, LD, FADA, CNSC, Principal Investigator — Baylor Health Care System
Locations (1):
- Baylor University Medical Center, Dallas, Texas, United States

REFERENCES:
- [Derived] Hasse JM, van Zyl JS, Felius J, Lima B, Jamil AK, Alam A. Bioimpedance Spectroscopy in Heart Transplantation: Posttransplant Changes in Body Composition and Effects in Outcomes. Transplantation. 2023 Nov 1;107(11):e305-e317. doi: 10.1097/TP.0000000000004678. Epub 2023 Jun 9. PMID 37291721